CLINICAL TRIAL: NCT05635630
Title: Predictive Value of Circulating Tumor DNA (ctDNA) for no Evidence of Disease (NED) Status in Metastatic Colorectal Cancer (mCRC) and Its Utility in Guiding Therapeutic Intervention: an Open-label, Prospective, Phase II Cohort Study
Brief Title: Predictive Value of ctDNA for NED Status in mCRC and Its Utility in Guiding Therapeutic Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Junjie Peng, MD, PhD, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ctDNA-nedCRC
Record Dates: First submitted 2022-11-03; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Colorectal Cancer; No Evidence of Disease Status; ctDNA Monitoring
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Circulating Tumor DNA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA positive (Experimental)
  Interventions: Other: ctDNA and adjuvant therapy
- ctDNA negative (Experimental)
  Interventions: Other: ctDNA

INTERVENTIONS:
Other: ctDNA and adjuvant therapy — Patients of ctDNA positive group receive individual adjuvant chemotherapy. The ctDNA status are evaluated every 2 months.
  Arms: ctDNA positive
Other: ctDNA — Patients of ctDNA negative group are monitored by ctDNA every 3 months.
  Arms: ctDNA negative

SUMMARY:
The goal of this clinical trial is to detect the prognostic value of longitudinal monitoring circulating tumor DNA (ctDNA) for no evidence of disease (NED) status in metastatic colorectal cancer (mCRC) patients and its utility in guiding therapeutic intervention. The main questions it aims to answer are:

1. Whether ctDNA monitoring could evaluate NED status ahead of normal radiologic monitoring. What about the concordance of evaluating NED status by ctDNA monitoring compared with normal radiologic monitoring?
2. Whether the patients with ctDNA positive status could benefit from early therapeutic intervention.

Patients who receive any kinds of therapies with the aim of NED and are confirmed by clinical and radiologic examination will go through longitudinal ctDNA monitoring. According to the results of ctDNA monitoring, the patients will be divided into ctDNA positive group and ctDNA negative group. Patients in ctDNA positive group will receive individual therapeutic plan decided by the investigator. Patients in ctDNA negative group will receive regular examinations. When radiologic recurrences are confirmed, the patients will be re-evaluated for a second opportunity of radical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old. Both male and female are eligible.
2. Late stage metastatic colorectal adenocarcinoma diagnosed by histology or cytology.
3. With potential opportunity of achieving NED status (including liver metastasis, lung metastasis, solitary lymph node metastasis, ovarian metastasis or focal pelvic metastasis), regardless of neo-adjuvant therapy or transforming therapy.
4. Patients who are intended for focal therapy, radical surgery, focal radiotherapy, radiofrequency ablation or interventional therapy (anhydrous alcohol injection or cryotherapy)
5. Eastern Cooperative Oncology Group (ECOG) grade 1-2.
6. Approve the informed consent.
7. Available for tumor sample obtained by resection or aspiration.
8. Available for peripheral blood collection (10mL per tube for 2 tubes)

Exclusion Criteria:

1. Cannot get histologic or cytologic diagnosis.
2. Clinical tumor, node, and metastasis (cTNM) stage I-III according to the American Joint Committee on Cancer (AJCC), the 8th edition.
3. Accompany with widespread metastasis and cannot achieve NED status by focal therapy, such as bone metastasis, peritoneum metastasis, diffuse liver or lung metastasis or malignant effusion, etc.
4. Inadequate bone marrow reserve and organ function.
5. Uncontrolled or severe systemic diseases, such as uncontrolled hyperplasia, severe infection, hepatitic B virus (HBV) infection, hepatitis C virus (HCV) infection, human immunodeficiency virus (HIV) infection, etc.
6. History of alcohol or drug abuse.
7. Pregnant or lactating women.
8. Cannot get tumor sample.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) time | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  To detect the RFS time in metastatic colorectal cancer (mCRC) patients with no evidence of disease (NED) status who received circulating tumor DNA (ctDNA) guided therapies.

SECONDARY OUTCOMES:
Overall survival (OS) time | From the date of surgery until the date of death from any cause, assessed up to 2 years.
  To detect the OS time in mCRC patients with NED status who received ctDNA guided therapies.
The positive rate of ctDNA in mCRC patients with NED status. | Post-operation 1 month
  When the NED status is confirmed by radiology post-operation, it will also be assessed the ctDNA positive rate.
The concordance index of ctDNA defined NED and radiology defined NED status. | When the clinic trail is finished, up to 2 years.
  In this study, we aim to evaluate the NED status by ctDNA and traditional radiologic methods. The concordance index will be used to detect the identity of two methods.
The rate of achieving NED status when relapses happen. | When the relapses happen, up to 2 years.
  When the diseases relapse during the follow-up. The multi-disciplinary treatment (MDT) team will discuss the opportunities to achieve a second NED status.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China